CLINICAL TRIAL: NCT04310488
Title: Assessment of Effects of Museum Prescription of A Montreal Museum Of Fine Arts Visit Tour in Primary Care Patients: a Cross-Sectional Study
Brief Title: Assessment of Effects of Museum Prescription of A Montreal Museum of Fine Arts Visit Tour in Primary Care Patients
Status: Withdrawn | Type: Observational
Why Stopped: PI has changed of institution. Project will be declare on the new institution ClinicalTrials.gov affiliation.
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Professor of Geriatrics, Holder of the Dr. Joseph Kaufmann Chair in Geriatric Medicine Clinician Scientist, Department of Medicine, Division of Geriatric Medicine Director of Centre of Excellence on Longevity, RUISSS McGill, McGill University, Jewish General Hospital
Other Study IDs: 2020-2091
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Museum; Mental Health; Quality of Life; Health, Subjective
Keywords: Museum; Art
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Centre of excellence self-administered (CESAM) questionnaire items — Complete a self-administered questionnaire within two days of their museum visit.

SUMMARY:
The objective of this study is to examine effects on mental and physical health and quality of life in primary care patients visiting the Montreal Museum of Fine Arts (MMFA), this visit being prescribed by their physician. To visit the MMFA and to complete after this visit a series of self-administered questionnaires within the two days after their visit at the museum

DETAILED DESCRIPTION:
During the past decade, museums have become involved in the care of patients by using art to improve their quality of life and well-being. Museums have, thus, emerged as new partners in public health. Very few programs developed by museums have focused on primary care patients who are a target audience for museum health program preventions. For the development of appropriate museum programs based on visit tour, there is a need to improve knowledge the effects of a museum visit prescribed by a primary care physician in patients. The objective of this study is to examine effects on mental and physical health and quality of life in primary care patients visiting the Montreal Museum of Fine Arts (MMFA), this visit being prescribed by their physician. Based on a cross-sectional study it will be prescribed to all patients consulting their primary care physician to visit the MMFA and to complete after this visit a series of self-administered questionnaires within the two days after their visit at the museum. The period of recruitment will be one year. The outcomes are the scores of the different questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Home Internet access with an electronic device (computer, pad or cellular phone)
3. Patient without dementia
4. Speak the language of the recruitment centre (French or English)

Exclusion Criteria:

1. dementia
2. participation refusal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Montreal Museum of Fine Arts visitors
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-13 (Estimated); Study Completion 2025-03-13 (Estimated)

PRIMARY OUTCOMES:
Socio-demographic characteristics from the primary care physician questionnaire | 1 day
  Primary care physician questionnaire is composed of 12 items exploring socio demographic items (age, gender), the reason perceived by the participants of the prescription and the effects of the visit on a scale form 0 (not at all) to 10 (extremely)
Mental health condition from the primary care physician questionnaire | 1 day
  Primary care physician questionnaire is composed of 12 items exploring socio demographic items (age, gender), the reason perceived by the participants of the prescription and the effects of the visit on a scale form 0 (not at all) to 10 (extremely)
Physical health condition | 1 day
  The Centre of excellence self-administered (CESAM) questionnaire items

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided